CLINICAL TRIAL: NCT02050711
Title: Effects of Pulmonary Rehabilitation on Computerized Respiratory Sounds in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Pulmonary Rehabilitation on Respiratory Sounds in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Alda Sofia Pires de Dias Marques, Senior Lecturer, Aveiro University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SFRH/BD/84665/2012
Record Dates: First submitted 2014-01-28; First posted 2014-01-31 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic obstructive pulmonary disease (COPD); Pulmonary rehabilitation; Computerized respiratory sounds
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Other): Patients will receive usual care from their general practitioners/pulmonologists.
  Interventions: Other: Usual care
- Pulmonary rehabilitation (Experimental): Patients will enrol in a 12-week PR program consisting on exercise training (3 times a week) and psychoeducation (once a week).
  Interventions: Behavioral: Pulmonary rehabilitation

INTERVENTIONS:
Behavioral: Pulmonary rehabilitation
  Arms: Pulmonary rehabilitation
Other: Usual care
  Arms: Usual care

SUMMARY:
The effect of pulmonary rehabilitation in patients with chronic obstructive pulmonary disease (COPD) has been based on systemic outcome measures, however, little is known about the effectiveness of this intervention on patients' lung function. The forced expiratory volume in one second (FEV1), despite of being the gold standard for assessing lung function in COPD, is poorly responsive to pulmonary rehabilitation. Thus, an objective and responsive outcome measure to assess the effect of pulmonary rehabilitation on lung function is needed.

Computerized respiratory sounds have been found to be a more sensitive indicator, detecting and characterizing the severity of respiratory diseases before any other measure, however its potential to detect changes after pulmonary rehabilitation has never been explored. Therefore, this study aims to assess the effects of pulmonary rehabilitation on the characteristics of computerized respiratory sounds in patients with COPD.

A randomized controlled study with one group undergoing pulmonary rehabilitation (n=25) and other group receiving standard care (n=25) will be conducted. The pulmonary rehabilitation program will included exercise training (3*week) and psychoeducation (1*week).

Computerized respiratory sounds, lung function, exercise capacity, quadriceps muscle strength, health-related quality of life and health services use will be assessed in both groups, at baseline, immediately post-intervention and at follow-ups (3 and 6 months after PR).

Descriptive and inferential statistics will be used.

It is expected that significant changes occur on the characteristics of computerized respiratory sounds in patients enrolled in the pulmonary rehabilitation group, in comparison with patients receiving standard care. Thus, computerized respiratory sounds could provide a simple, objective and non-invasive measure to assess lung function changes after pulmonary rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of COPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria;
* ≥ 18 years old;
* clinical stability for 1 month prior to the study (no hospital admissions, exacerbations or changes in medication);
* able to provide their own informed consent.

Exclusion Criteria:

* presence of concomitant respiratory diseases;
* presence of severe psychiatric conditions;
* presence of severe neurologic/ musculoskeletal conditions and/or unstable cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2013-03-20 (Actual); Study Completion 2013-09-30 (Actual)

PRIMARY OUTCOMES:
Change in respiratory sounds | 1 week prior intervention; 1, 12 and 24 weeks post intervention
  Computerized respiratory sounds will be recorded with modified stethoscopes at seven chest locations: trachea; posterior right and left; anterior right and left and lateral right and left, as recommended by the Computerized Respiratory Sound Analysis (CORSA) guidelines.

SECONDARY OUTCOMES:
Change in lung function | 1 week prior intervention; 1, 12 and 24 weeks post intervention
  Lung function will be assessed with a spirometric test, following the American Thoracic Society/European Respiratory Society guidelines.
Change in exercise capacity | 1 week prior intervention; 1, 12 and 24 weeks post intervention
  Exercise capacity will be assessed with the 6-minute walk test, following the American Thoracic Society guidelines.
Change in quadriceps muscle strength | 1 week prior intervention; 1, 12 and 24 weeks post intervention
  Quadriceps isotonic muscle strength will be assessed with the 1 repetition maximum (1-RM), following the American College of Sports Medicine guidelines.
Change in health-related quality of life | 1 week prior intervention; 1, 12 and 24 weeks post intervention
  The St. George's Respiratory Questionnaire (SGRQ) is a disease-specific instrument designed to measure quality of life in patients with chronic lung disease. It has 3 domains: symptoms, activities and impact. Scores range from 0 to 100 and higher values indicate poorer quality of life.
Change in health services use | 1 week prior intervention; 1, 12 and 24 weeks post intervention
  number of visits to casualty; number and duration of hospital admissions.

CONTACTS AND LOCATIONS:
Overall Officials: Alda S Marques, PhD, Principal Investigator — School of Health Sciences of the University of Aveiro (ESSUA)
Locations (1):
- University of Aveiro, Aveiro, Portugal

REFERENCES:
- [Background] Marques A, Oliveira A, Jacome C. Computerized adventitious respiratory sounds as outcome measures for respiratory therapy: a systematic review. Respir Care. 2014 May;59(5):765-76. doi: 10.4187/respcare.02765. Epub 2013 Sep 17. PMID 24046460
- [Background] Jacome C, Marques A. Pulmonary rehabilitation for mild COPD: a systematic review. Respir Care. 2014 Apr;59(4):588-94. doi: 10.4187/respcare.02742. Epub 2013 Oct 8. PMID 24106321